CLINICAL TRIAL: NCT00128089
Title: Phase 1 Trial of A New Dietary Treatment of Obesity Related Type 2 Diabetes
Brief Title: Trial of New Dietary Treatment of Diabetes
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Manassas Internal Medicine (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-1
Record Dates: First submitted 2005-08-08; First posted 2005-08-09 (Estimated); Last update posted 2005-12-21 (Estimated); Status verified 2005-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Obesity; Dietary treatment; Fasting as medical therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

INTERVENTIONS:
Behavioral: Dietary treatment

SUMMARY:
This is a preliminary trial of a new dietary approach to the treatment of obesity related type 2 diabetes.

Study terminated December 19, 2005 for administrative reasons.

DETAILED DESCRIPTION:
Traditional dietary treatment of type 2 diabetes is complicated and often fails.

This is a dietary treatment that uses fingerstick testing of blood sugars and a remarkably simple algorithm to promptly lower the blood glucose to treatment goals.

A series of 10 overweight type 2 diabetic patients not well controlled, or needing medication for control, will be recruited to follow this plan; followup is to be until 6 months after the last patient is enrolled, or when all patients have normal A1Cs with no medication, whichever comes first.

Primary endpoints to be measured are A1C, weight loss (in pounds and BMI reduction) and medication reduction. Secondary endpoints are occurrences of hypoglycemia, reduction of medications for hypertension and hyperlipidemia, and patient satisfaction. As this is a Phase 1 trial, the only control group is historical controls (the patients themselves and the medical literature).

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus, type 2
* Obesity
* Ability to attend office visits in Manassas, Virginia

Exclusion Criteria:

* Dementia
* Institutionalized living
* Retinopathy, neuropathy
* Pregnancy
* Serious health problems such as heart disease or stroke

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2005-08; Study Completion 2005-12

PRIMARY OUTCOMES:
Glycated hemoglobin (A1C) changes
Weight (body mass index [BMI]) loss
Diabetes medication reduction

SECONDARY OUTCOMES:
Hypoglycemia
Other medication reduction
Patient satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: John F Cary, MD, Principal Investigator — Manassas Internal Medicine
Locations (1):
- Manassas Internal Medicine, Manassas, Virginia, United States